CLINICAL TRIAL: NCT00116376
Title: A Phase I/II, Two-arm, Multicenter, Dose Escalation Study of Oral AEE788 Administered on a Continuous Once Daily Dosing Schedule in Adult Patients With Recurrent or Relapsing Glioblastoma Multiforme
Brief Title: Study of AEE788 in Patients With Recurrent/Relapse Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEE788A2103; NCT00085215 (obsolete NCT alias)
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; recurrent/relapse; EGFR; VEGFR
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — AEE 788

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AEE788 + non EIACD (Experimental)
  Interventions: Drug: AEE788
- AEE788 + EIACD (Experimental)
  Interventions: Drug: AEE788

INTERVENTIONS:
Drug: AEE788

SUMMARY:
AEE788 is an orally active, reversible, small-molecule, multi-targeted kinase inhibitor with potent inhibitory activity against the ErbB and VEGF receptor family of tyrosine kinases. It has an IC50 of less than 100 nM against p-EGFR, p-ErbB2, and p-KDR (VEGFR2). This study will assess the safety, pharmacokinetic/pharmacodynamic (PK/PD) profiles and clinical activity of AEE788 in a recurrent GBM population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM in first or second recurrence or relapse
* Adequate hematologic, hepatic and renal function
* Age ≥ 18 years
* Karnofsky performance status score ≥ 70%
* Life expectancy ≥ 12 weeks

Exclusion Criteria:

* Peripheral neuropathy > grade 1
* Diarrhea > grade 1
* Gastrointestinal dysfunction
* Compromised cardiac function
* Concurrent severe and/or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 years
Dose limiting toxicity | 2 years

SECONDARY OUTCOMES:
Safety, tolerability, pharmacokinetic profiles, change in plasma markers of angiogenesis, tumor PK levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, MD, Principal Investigator — Duke University; Charles Conrad, MD, Principal Investigator — M.D. Anderson Cancer Center; Timothy Cloughesy, MD, Principal Investigator — University of California, Los Angeles; Michael Prados, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California at Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - The Brain Tumor Center at Duke, Duke University Medical Center, Box 3624 Dumc, Trent Drive, Durham, North Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas